CLINICAL TRIAL: NCT04991376
Title: Differentiation of Acute Kidney Injury in Sepsis and Due to Nephrotoxic Antibiotic Treatment With Vancomycin and Gentamicin Based on Measurements of Specific miRNAs
Brief Title: Specific miRNAs in Sepsis and Nephrotoxic Antibiotic Treatment
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Collaborators: Palacky University (Other); University Hospital Olomouc (Other); University of Ostrava (Other); Technical University of Ostrava (Unknown)
Responsible Party: Sponsor
Other Study IDs: IK-01-miRNA; 01 - RVO - FNOs/2019 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2021-07-27; First posted 2021-08-05 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Sepsis; Septic Shock; Acute Kidney Injury
Keywords: sepsis; septic shock; acute kidney injury; microRNA; nephrotoxicity; vancomycin; gentamicin
MeSH Terms: conditions — Sepsis; Shock, Septic; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vancomycin: Critically ill patients who suffered from sepsis, treated with vancomycin.
  Interventions: Diagnostic Test: Blood-specific miRNA levels
- Gentamicin: Critically ill patients who suffered from sepsis, treated with gentamicin.
  Interventions: Diagnostic Test: Blood-specific miRNA levels
- Other antibiotic groups: Critically ill patients who suffered from sepsis, treated by other antibiotic groups except for vancomycin or aminoglycoside (gentamicin).
  Interventions: Diagnostic Test: Blood-specific miRNA levels

INTERVENTIONS:
Diagnostic Test: Blood-specific miRNA levels — Blood-specific miRNA levels associated with renal tubular damage change in patients treated with vancomycin or gentamicin compared to septic patients treated with other antimicrobials.

SUMMARY:
Critically ill patients are prone to develop acute kidney injury due to sepsis itself and by administration of potentially nephrotoxic antibiotic treatment (vancomycin or gentamicin). Blood-specific miRNA levels associated with renal tubular damage change in patients treated with vancomycin or gentamicin compared to septic patients treated with other antimicrobials.

DETAILED DESCRIPTION:
Sepsis is generally defined as a life-threatening and dysregulated reaction to infection (bacterial, fungal, or viral) leading to systemic inflammation and organ dysfunction including acute kidney injury [1]. Acute kidney injury in critically ill patients is a common and usually serious condition associated with increased patient morbidity and mortality. Critically ill patients are prone to develop acute kidney injury due to sepsis itself and by administration of potentially nephrotoxic antibiotic treatment (vancomycin or aminoglycoside-gentamicin). To prevent nephrotoxicity and avoid subtherapeutic dosing, drug serum concentrations are usually monitored, with adjustment of dose or dosing interval according to the pharmacokinetic model. However, renal tubular injury can occur even if the treatment is optimally set. In the quest for new preventive or therapeutic targets (biomarkers) in septic/nephrotoxic acute renal damage, a current research focus in microRNAs. Based on data from previously published experimental and human studies we identified specific miRNAs associated with biochemical pathways involved in inflammation, organ ischemia, and nephrotoxicity with their exact determination and time-changing detection during the seven days in studied patients. Blood-specific miRNA levels associated with renal tubular damage change in patients treated with vancomycin or gentamicin compared to septic patients treated with other antimicrobials.

Sampling method:

Whole blood samples were taken on the first, fourth, and seventh days of antibiotic treatment. The first 24 samples (8 patients) were extracted in duplicate for screening of the selected miRNAs. Blood samples were collected into 2.5 mL tubes (Vacutainer® PAXgene, PreAnalytiX® GmbH, A Qiagen/BD Company, Switzerland). Concomitant-ly, the blood samples for NGAL determination were collected into 2.6 or 2 mL neutral tubes (S-Monovette® K3 EDTA, 2.6 mL, red, Sartstedt AG & Co. KG, Germany; or Vacuette® K3 EDTA 2 mL, violet, Greiner Bio-One GmbH, Germany). The blood samples for biochemical (renal and inflammatory) parameters (serum creatinine, interleukin-6, procalcitonin, C-reactive protein) were collected concomitantly with other dai-ly routine biochemical parameters (S-Monovette® serum-gel, 4.9 mL, brown, Sartstedt AG & Co. KG, Germany in University Hospital Ostrava; or Vacuette® serum-gel, 5.0 mL, red, Greiner Bio-One GmbH, Germany in University Hospital Olomouc). The serum antibiotic concentrations (vancomycin and gentamicin) were monitored according to standard care in both cooperating hospitals without needing more blood samples for study.

ELIGIBILITY:
Inclusion Criteria:

- Critically ill adult septic patients with or without acute kidney injury treated by antimicrobial therapy

Exclusion Criteria:

- Patients in the chronic dialysis program, with stage 4 and 5 chronic kidney disease, or concomitantly treated with another potentially severe nephrotoxic medication (cisplatin, colistin) or combination vancomycin/gentamicin.

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Critically ill patients suffering from sepsis and treated with vancomycin, gentamicin, or other antibiotic groups.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
miRNAs expression over 7 days of treatment | 7 days
  Determine and investigate specific circulating miRNAs linked to sepsis itself, septic, ischemic, or nephrotoxic acute kidney injury in patients suffered from sepsis. Tracking changes in miRNAs expression over 7 days of treatment with nephrotoxic (vancomycin or gentamicin) as compared with other, non-nephrotoxic antibiotic treatment.

SECONDARY OUTCOMES:
Association between circulating miRNA expression and serum neutrophil gelatinase-associated lipocalin (NGAL) and other renal or inflammatory markers | 7 days
  Association between circulating miRNA expression and serum neutrophil gelatinase-associated lipocalin (NGAL) and other renal or inflammatory markers to assess the potential of these small RNAs as pathophysiological biomarkers of nephrotoxic acute kidney injury or preventive, or therapeutic targets in sepsis and/or acute kidney injury.

CONTACTS AND LOCATIONS:
Overall Officials: Naděžda Petejová, Assoc.Prof.,MD,PhD,MSc, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Eckardt KU, Kasiske BL. Kidney disease: improving global outcomes. Nat Rev Nephrol. 2009 Nov;5(11):650-7. doi: 10.1038/nrneph.2009.153. Epub 2009 Sep 29. PMID 19786993
- [Background] Petejova N, Martinek A, Zadrazil J, Kanova M, Klementa V, Sigutova R, Kacirova I, Hrabovsky V, Svagera Z, Stejskal D. Acute Kidney Injury in Septic Patients Treated by Selected Nephrotoxic Antibiotic Agents-Pathophysiology and Biomarkers-A Review. Int J Mol Sci. 2020 Sep 26;21(19):7115. doi: 10.3390/ijms21197115. PMID 32993185
- [Derived] Petejova N, Martinek A, Zadrazil J, Klementa V, Pribylova L, Bris R, Kanova M, Sigutova R, Kacirova I, Svagera Z, Bace E, Stejskal D. Expression and 7-day time course of circulating microRNAs in septic patients treated with nephrotoxic antibiotic agents. BMC Nephrol. 2022 Mar 19;23(1):111. doi: 10.1186/s12882-022-02726-6. PMID 35305556